CLINICAL TRIAL: NCT00001168
Title: Teaching Protocol for the Evaluation of Plasma Lipoproteins
Brief Title: Evaluation of Lipoproteins
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 790100; 79-H-0100
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-08-19

CONDITIONS: Evaluation of Plasma Lipoproteins
Keywords: High Cholesterol; High HDL; Low HDL; LCAT Defiency; Natural History; Type III Hyperlipoproteinemia; Plasma Lipoproteins
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipoproteinemia Type III

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dyslipidemia: Dyslipidemia
  Interventions: Behavioral: Balanced diet

INTERVENTIONS:
Behavioral: Balanced diet — Dietary studies for the diagnosis of post-prandial hyperlipidemia will include a 3 week period while subjects are on a baseline, isoweight, 15% fat, 42% carbohydrate, normal polyunsaturated fat ratio (0.1-0.3) 250-300 mg cholesterol diet.

SUMMARY:
Lipoproteins are particles that carry fats such as cholesterol and triglycerides through the blood stream. These particles are involved in causing blood vessel disease that can lead to conditions like hardening of the arteries (atherosclerosis) or heart attacks (myocardial infarctions).

This study is designed to look closely at the factors affecting lipoproteins. Researchers plan to study patients and normal volunteers by measuring lipoprotein levels in the blood. Patients and volunteers will be placed on a balanced diet during the study. In addition, researchers plan to measure levels of various hormone and enzymes in the blood. Patients and volunteers participating in the study may be asked to undergo more specific tests in order to collect more information about lipoprotein metabolism.

This study may not provide direct benefits to patients and volunteers participating in it. However, information gathered from this study may help researchers develop better skills and techniques to diagnose and treat patients with diseases of lipoprotein metabolism.

DETAILED DESCRIPTION:
The lipoprotein transport system is vital to the delivery of the hydrophobic fats that are carried in the aqueous environment of the blood. The lipoprotein particles that comprise this system are polydisperse and contain triglycerides, free and esterified cholesterol, phospholipids and proteins. Inborn errors in the lipoprotein transport system lead to alterations in both the steady state concentrations of the various lipoproteins and in the metabolism of these particles. These inborn errors lead to both hyperlipoproteinemia and hypolipoproteinemia. Profound changes in the ambient lipoprotein concentrations have a variety of clinical manifestations. The present study protocol is designed to permit a full evaluation of the lipids, lipoproteins, and apolipoproteins, in patients with potential genetic defects in these processes. The protocol will also permit training of students, staff clinicians, physician assistants, nurse practitioners, dieticians and post-doctoral fellows in the evaluation and treatment of patients with dyslipidemias. The study population will include patients which are referred to the Lipid Service from private care providers, academic institutions, or the NHLBI Lipid website, with any of the following potential lipid abnormalities or clinical stigmata associated with dyslipoproteinemias: a) increased plasma levels of cholesterol, triglycerides, HDL-cholesterol or LDL-cholesterol b) decreased plasma concentrations of cholesterol and HDL-cholesterol c) postprandial hyperlipidemia or d) eruptive xanthomas, xanthelasma, tuberous or tendinous xanthomas, or corneal opacities.

ELIGIBILITY:
* INCLUSION CRITERIA:

The following is a representative list of the types of patient presentations and potential diagnoses eligible for this protocol:

Plasma cholesterol levels greater than 200 mg/dl or less than 120 mg/dl - includes patients with diagnoses such as familial hypercholesterolemia, familial combined hyperlipidemia, sitosterolemia, cholesteryl ester storage disease, Erdheim chester disease, lipoprotein lipase, hepatic lipase or apo-CII deficiency, and dysbetalipoproteinemia.

Plasma LDL-C levels greater than 130 mg/dl or less than 70 mg/dl - includes patients with diagnoses such as familial hypercholesterolemia, familial combined hyperlipidemia, lipoprotein lipase, hepatic lipase, or apo-CII deficiency, sitosterolemia, dysbetalipoproteinemia, abetalipoproteinemia and hypobetalipoproteinemia.

Plasma HDL-C levels greater than 70 mg/dl or less than 25 mg/dl - includes patients with deficiency of cholesteryl ester transfer protein, lecithin cholesterol acyltransferase, phospholipid transfer protein, lipoprotein lipase, hepatic lipase, or apo-CII, and Tangier disease.

Plasma triglyceride levels greater than 150 mg/dl - includes patients with deficiency of lipoprotein lipase, hepatic lipase or apoC-II, dysbetalipoproteinemia, Type IV and Type V hyperlipidemia.

EXCLUSION CRITERIA:

Inability to provide informed consent.

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: unlimited
Sampling Method: Non-Probability Sample
Enrollment: 1017 (Actual)
Dates: Start 1979-01-01 (Actual)

PRIMARY OUTCOMES:
Screening and evaluation of individuals with potential disorders of lipid metabolism in order to provide training for professional Lipid Service staff in the evaluation and treatment of patients with genetic dyslipoproteinemias. | Six years
  Training for professional Lipid Service staff in the evaluation and treatment of patients with genetic dyslipoproteinemias

SECONDARY OUTCOMES:
Some of these patients may be candidates for enrollment in other Lipid Service research protocols. | six years
  Some of these patients may be candidates for enrollment in other Lipid Service research protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Shamburek, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1979-H-0100.html